CLINICAL TRIAL: NCT05422586
Title: Validation Study of Penn's Way to Drive Telematics Research Application
Brief Title: Way To Drive Validation Study
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, M. Kit Delgado, MD, Assistant Professor of Emergency Medicine, University of Pennsylvania
Other Study IDs: 849755
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Validity; Distracted Driving; Driving Behaviors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Way to Drive is a smart phone-based driving telematics application. Research participants are invited to download the app, which uses phone sensors to track driving behaviors including mileage, hard breaking events, and handheld phone use while driving, measured as the phone screen being unlocked while the phone is in the hand and the vehicle is in motion. Before the study team launches a clinical trial using the app, the researchers will test its capabilities and reliability.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older (only adult drivers will be invited)
* Willing to download Way to Drive and allow it to track the user's location while the user is in motion (i.e. over 5mph)
* Will make at least 4 driving trips per week for the duration of the study.
* Able to provide informed consent

Exclusion Criteria:

* Under 18 Cannot complete online surveys
* Does not have smart phone
* Not willing to download Way to Drive app and allow location tracking while in motion
* Will not be driving at least 4 times per week during the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults who completed in the study team's recent clinical trial with User Based Insurance customers and stated interest in being contacted about further research opportunities. The adults participated in a driving monitoring study (May 2021) and met the eligibility criteria, including 4 trips per week.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2022-07-17 (Actual); Primary Completion 2022-08-13 (Actual); Study Completion 2022-08-13 (Actual)

PRIMARY OUTCOMES:
Number of driving trips classified correctly (driver/passenger) by the Way to Drive Telematics App | 28 days
  Measured by the driving and behavior when the car is in motion by the Way to Drive app.

SECONDARY OUTCOMES:
Number of driving events accurately captured (trip captured or missing) by Way to Drive Telematics App | 28 days
  Measured using phone sensor data to detect when the vehicle is in motion.

CONTACTS AND LOCATIONS:
Overall Officials: Mucio Delgado, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be made available to other researchers upon request.
Supporting Information: SAP
Time Frame: Data will be made 5 weeks after request and indefinitely thereafter.